CLINICAL TRIAL: NCT02661074
Title: Protists and Nematodes Fish Parasites: From Their Circulation in Ecosystems to Their Impact on Human Health - Prevalence of Fish Allergy in Occupational Settings.
Brief Title: Anisakis Blastocystis Cryptosporidium Fish Prevalence
Acronym: ABCFish1
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut Pasteur de Lille (Other); ANSES (Other); Région Nord-Pas de Calais, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_42; 2014-A00853-44 (Other: ID RCB number, ANSM)
Record Dates: First submitted 2016-01-13; First posted 2016-01-22 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Anisakis; Allergy; Occupational Exposure
Keywords: Fisherman; Fish industry
MeSH Terms: conditions — Anisakiasis; Hypersensitivity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Fishermen: Fisherman followed by the "Service de Santé des Gens de Mer" of Boulogne-sur-Mer, France (occupational exposure to fish).
  A questionnaire will be completed.
  Interventions: Other: Questionnaire
- Fish processing factories: Workers of fish processing factories who are followed by the "Service de Santé au Travail" (ASTIL) of Boulogne-sur-Mer, France (occupational exposure to fish).
  A questionnaire will be completed.
  Interventions: Other: Questionnaire
- Control: Workers who are followed by the "Service de Santé au Travail" (ASTIL) of Boulogne-sur-Mer, France, but do not work in fish processing factories.
  A questionnaire will be completed.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire will be completed in order to collect data on:
  * Potential allergic manifestations after fish contact: asthma, allergic rhinitis, conjunctivitis, chronic or acute urticaria, dermatitis/eczema, or severe allergic manifestations (angioedema, bronchospasm, anaphylaxis),
  * Occupational and/or domestic exposure to fish.

SUMMARY:
Anisakidae frequently infect fish species that are commonly eaten by humans. Some of them are recognized as zoonotic agents, and have a high impact on human health.

Infestation results from the ingestion of living larvae from contaminated fishes. It can be asymptomatic or symptomatic, resulting in acute gastric, acute intestinal or chronic forms. Allergic manifestations are frequently encountered in gastric forms, but isolated allergic symptoms can occur after ingestion of Anisakidae antigens in raw or cooked fish. Cutaneous contact or Anisakis allergen inhalation have also been reported to induce allergy/anaphylactic reactions or sensitization in the occupational setting in Spain, Italy, Sicilia or South Africa. But no data is available in France.

In this context, the investigators propose to determine and compare the frequency and characteristics of fish allergy in fish workers (fishermen and fish-processing factory workers) and a control population of workers without occupational exposure to fish, in Boulogne-sur-Mer, which is an important fishing port in France, and the first European center for fish processing.

DETAILED DESCRIPTION:
162 fishermen, 162 fish-processing factory workers, and 162 control subjects will be consecutively recruited by their occupational doctor during a routine consultation. A standardized questionnaire will be used to collect epidemiological and clinical data on potential allergic manifestation resulting from digestive, cutaneous, or respiratory contact with fish. Domestic and occupational risk factors for fish and Anisakis exposure will also be collected for both allergic and non-allergic patients.

ELIGIBILITY:
Inclusion Criteria:

* Fisherman followed by the "Service de Santé des Gens de Mer" of Boulogne-sur-Mer, fish-processing factory worker followed by the "Service de Santé au Travail" of Boulogne-sur-Mer, or worker followed by the "Service de Santé au Travail" of Boulogne-sur-Mer, but not working in a fish-processing factory.

Exclusion Criteria:

* Pregnant or breast-feeding female
* Patient with no social insurance
* Patient unwilling to comply with the protocol
* Patient unable to understand the study and its objectives
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include the following 3 groups:
  * Fishermen followed by the "Service de Santé des Gens de Mer" of Boulogne-sur-Mer,
  * Fish-processing factory workers followed by the "Service de Santé au Travail" of Boulogne-sur-Mer,
  * A control group composed of workers followed by the "Service de Santé au Travail" of Boulogne-sur-Mer, but not working in a fish-processing factory.
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The prevalence of fish allergy | contact by phone during 30 min at only visit (inclusion)
  Difference in the prevalence of fish allergy between occupationally exposed (fishermen and fish-processing factory workers) and non-exposed subjects.
  the fish allergy is definied by clinical diagnosis based on the presence of clinical manifestations of allergy in contact with the fish ( APC)

SECONDARY OUTCOMES:
Frequencies history of infections Anisakis spp. | contact by phone during 30 min at only visit (inclusion)
  Comparison between occupationally exposed ( E: fishermen and fish-processing factory workers) and non-exposed subjects(NE)
Frequency of fish allergies, history of infections Anisakis spp. (clinical diagnosis) | contact by phone during 30 min at only visit (inclusion)
  comparison between occupationally exposed and non-exposed subjects for previous Anisakidosis.
  Fish exposure will be determined taking into account the handled fish species and the local prevalences of fish parasites.
history of infections Anisakis spp. (clinical diagnosis) | contact by phone during 30 min at only visit (inclusion)
  comparison between occupationally exposed and non-exposed subjects for previous Anisakidosis.
  Fish exposure will be determined taking into account the handled fish species and the local prevalences of fish parasites.
Frequency of risk factors for occupational or domestic exposure to fish: | contact by phone during 30 min at only visit (inclusion)
  comparison subjects (i) allergic or non-allergic Fish (APC + APC-vs) (ii) with or without a history of infection Anisakis spp. (IA + vs IA-).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DUTOIT, MD, Principal Investigator — University Hospital, Lille
Locations (3):
- France (3):
  - Centre ASTIL, Boulogne-sur-Mer
  - Service de Santé des Gens de Mer, Boulogne-sur-Mer
  - CHRU, Lille

IPD SHARING:
Plan to Share IPD: No